CLINICAL TRIAL: NCT00503178
Title: Biological Imaging Guided Antalgic Radiotherapy of Bone Metastases (Phase II Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/098
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Bone Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing imaging guided radiotherapy. (Experimental)
  Interventions: Procedure: Biological imaging guided antalgic radiotherapy

INTERVENTIONS:
Procedure: Biological imaging guided antalgic radiotherapy — Biological imaging guided antalgic radiotherapy is followed.

SUMMARY:
Highly selective irradiation requires accurate target definition by high-resolution three-dimensional imaging. Co-registration of FDG-PET and high-resolution CT might be the imaging modality of choice. This choice might target radiation therapy precisely to the intra-osseous volume that is responsible for pain and to spare selectively healthy bone in the vicinity of the metastasis. This strategy could result in equal anti-pain efficacy as conventional large volume radiotherapy, but could allow bone remodeling and preservation of bone structural strength in the vicinity and could lead to reduced toxicity to neighboring organs.

ELIGIBILITY:
Inclusion Criteria:

* Painful bone metastasis of solid tumors
* A maximum number of bone metastases less or equal to 3
* Life expectancy > 6 months
* Minimum age 21 years
* Signed informed consent

Exclusion Criteria:

* Previous radiotherapy to the painful site
* Bone metastasis from malignant melanoma or renal cell carcinoma
* Associated fracture or extra-osseous component

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

PRIMARY OUTCOMES:
Pain assessment | t0

SECONDARY OUTCOMES:
Acute toxicity | t0
Bone remodeling | t0
Resulting volumes of the targets and functional active areas | t0
Mismatch and/or overlap areas | t0

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be